CLINICAL TRIAL: NCT03972176
Title: Determination of Perinatal Exposure to Non-caloric Sweeteners. Implications for the Development of Preferences for Sweet Taste, and Weight Gain During the First Year of Life
Brief Title: Impact of Perinatal Exposure to Non-caloric Sweeteners on Food Preferences and Weight Gain in the First Year of Life
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Chile (Other)
Collaborators: University of Concepcion, Chile (Other); Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Responsible Party: Principal Investigator, Martin Gotteland, Head, Lab. of Digestive Physiology, University of Chile
Other Study IDs: UChile-Fonis SA18I0062
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Exposures Associated With Pregnancy, Delivery and Lactation
Keywords: non-caloric sweetener; Amniotic liquid; Breastmilk; Infant gain weight; Sweet taste preferences; Taste receptor polymorphism; Breastmilk microbiota; Infant gut microbiota; Salivary insulin
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During last years, non-caloric sweeteners (NCSs) have been increasingly incorporated into foodstuffs in replacement of sucrose in Chile. This situation has reached a point where it is currently difficult to find sugary foods without NCSs. As a result, the voluntary and involuntary consumption of these additives is growing significantly in the population, increasing the risk of exceeding the acceptable daily intake (ADI), especially for children. This situation is worrying as recent evidence suggests that NCSs are not inert in the body and can trigger adverse metabolic effects. For example, the consumption of beverages with NCSs has been shown to favor the development of obesity and type-2 diabetes in children and adults, and a recent study reported that the intake of NCSs during pregnancy was associated with a greater weight gain of the child at one year. It is likely that certain NCSs pass into the amniotic fluid and that the fetus is exposed to some of these compounds during pregnancy. This situation would persist in the infant through breast milk, as some studies detected sucralose and acesulfame-K in this fluid, even in mothers who claimed not to consume them. However, the real impact of NCS exposure during the neonatal period on the child health has been few studied. Therefore, the aim of this study is to determine the concentration of NCSs in samples of amniotic liquid and breastmilk and to correlate these data with the NCS intake by the mothers. Mothers/children will be classified in quintiles according to the results obtained. In the children from quintiles 1 and 5, we will also study whether neonatal exposure to NCSs may affect the sweet taste threshold and the preferences for this taste, the levels of salivary insulin and the weight gain in the first year. Breastmilk microbiota and child fecal microbiota will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Women with at least 36 weeks of gestation
* Spanish-speaking
* Elective cesarean delivery

Exclusion Criteria:

* Multiple pregnancy
* Type-2 diabetes
* Intelectual disability
* Presence of infectious disease compatible with chorio-amnionitis or immunosupression
* Newborns with serious pathologies affecting their growth

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 315 dyades mother/child recruited at the San Jose Hospital Maternity
Sampling Method: Probability Sample
Enrollment: 315 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Mothers with breastmilk NCSs | One month post-partum
  Proportion of mothers with detectable NCSs in their breastmilk

SECONDARY OUTCOMES:
Mothers with amniotic liquid NCSs | At delivery
  Proportion of mothers with detectable NCSs in their amniotic liquid
Consumption of NCSs by the mothers | At recruitment (in the last month of pregnancy) and at 1 mont post-partum
  Daily intake (mg/d) of sucralose, acesulfame-K, cyclamate, saccharin and stevia evaluated through a validated consumer trend survey
Pregnancy complications | At delivery
  Percentages of mothers with preclampsia, hypertension, gestacional diabetes, infections, or preterm labor
Breastmilk concentrations of NCSs | One month post-partum
  Concentrations of sucralose, acesulfame-K, cyclamate, saccharin, steviol in breastmilk samples
Amniotic liquid concentrations of NCSs | At delivery
  Concentrations of sucralose, acesulfame-K, cyclamate, saccharin, steviol in amniotic liquid samples
Sweet taste of breastmilk | One month post-partum
  Intensity (arbitrary units) of sweet taste in breast milk samples, as detected by e-tongue
Sweet taste of amniotic liquid | At delivery
  Intensity (arbitrary units) of sweet taste in amniotic liquid samples, as detected by e-tongue
Threshold of sweet taste in children | 6 months
  Determination of sweet taste threshold (lower concentration of sucrose detected) in children from quintiles 1 and 5 of classification according to the concentrations of NCS in breast milk that received
Food preferences in children | At 6 month of age
  Food consumption in children from quintiles 1 and 5 of classification according to the concentrations of NCS in breast milk that receiveded,through a validated consumer trend survey
Salivary insulin in children | 6 months
  Salivary concentration of insulin (pg/ml) in children from quintiles 1 and 5 of classification according to the concentrations of NCS in breast milk that they received
Infant gain weight | At 12 months
  Changes in weight (kg) during the first year of life
Breast milk microbiota diversity | At one month post-partum
  Intraindividual diversity of the breastmilk microbiota evaluated by Shannon index in samples from quintiles 1 and 5 of classification according to their NCS concentrations
Breast milk microbiota composition | At one month post-partum
  Relative abundancies of the different bacterial taxa from the breastmilk microbiota, detected by high throughput sequencing, in samples from quintiles 1 and 5 of classification according to their NCS concentrations
Fecal microbiota diversity in children | At six months post-partum
  Intraindividual diversity of the fecal microbiota, evaluated by Shannon index, in children from quintiles 1 and 5 of classification according to the concentrations of NCS in breast milk that they received
Fecal microbiota composition in children | At six months post-partum
  Relative abundancies of the different bacterial taxa from the fecal microbiota, detected by high throughput sequencing, in children from quintiles 1 and 5 of classification according to the concentrations of NCS in breast milk that they received
Polymorphism of sweet taste receptor in children | At six months post-partum
  Proportions of children presenting the different polymorphisms on the sweet taste receptor gene.

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Sambra, MaSc, Principal Investigator — University of Chile; Sandra Lopez, PhD, Principal Investigator — University of Chile; Paola Caceres, MaSc, Principal Investigator — University of Chile; Francisco Perez, PhD, Principal Investigator — University of Chile; Fabien Magne, PhD, Principal Investigator — University of Chile; Edgar Pastene, PhD, Principal Investigator — University of Concepción

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Popkin BM, Hawkes C. Sweetening of the global diet, particularly beverages: patterns, trends, and policy responses. Lancet Diabetes Endocrinol. 2016 Feb;4(2):174-86. doi: 10.1016/S2213-8587(15)00419-2. Epub 2015 Dec 2. PMID 26654575
- [Background] Brown RJ, de Banate MA, Rother KI. Artificial sweeteners: a systematic review of metabolic effects in youth. Int J Pediatr Obes. 2010 Aug;5(4):305-12. doi: 10.3109/17477160903497027. PMID 20078374
- [Background] Sylvetsky AC, Walter PJ, Garraffo HM, Robien K, Rother KI. Widespread sucralose exposure in a randomized clinical trial in healthy young adults. Am J Clin Nutr. 2017 Apr;105(4):820-823. doi: 10.3945/ajcn.116.144402. Epub 2017 Feb 22. PMID 28228424
- [Background] Duran Aguero S, Angarita Davila L, Escobar Contreras MC, Rojas Gomez D, de Assis Costa J. Noncaloric Sweeteners in Children: A Controversial Theme. Biomed Res Int. 2018 Jan 8;2018:4806534. doi: 10.1155/2018/4806534. eCollection 2018. PMID 29511682
- [Background] Sylvetsky A, Rother KI, Brown R. Artificial sweetener use among children: epidemiology, recommendations, metabolic outcomes, and future directions. Pediatr Clin North Am. 2011 Dec;58(6):1467-80, xi. doi: 10.1016/j.pcl.2011.09.007. Epub 2011 Oct 14. PMID 22093863
- [Background] Ruanpeng D, Thongprayoon C, Cheungpasitporn W, Harindhanavudhi T. Sugar and artificially sweetened beverages linked to obesity: a systematic review and meta-analysis. QJM. 2017 Aug 1;110(8):513-520. doi: 10.1093/qjmed/hcx068. PMID 28402535
- [Background] Burke MV, Small DM. Physiological mechanisms by which non-nutritive sweeteners may impact body weight and metabolism. Physiol Behav. 2015 Dec 1;152(Pt B):381-8. doi: 10.1016/j.physbeh.2015.05.036. Epub 2015 Jun 3. PMID 26048305
- [Background] Halldorsson TI, Strom M, Petersen SB, Olsen SF. Intake of artificially sweetened soft drinks and risk of preterm delivery: a prospective cohort study in 59,334 Danish pregnant women. Am J Clin Nutr. 2010 Sep;92(3):626-33. doi: 10.3945/ajcn.2009.28968. Epub 2010 Jun 30. PMID 20592133
- [Background] Rother KI, Sylvetsky AC, Schiffman SS. Non-nutritive sweeteners in breast milk: perspective on potential implications of recent findings. Arch Toxicol. 2015 Nov;89(11):2169-71. doi: 10.1007/s00204-015-1611-9. Epub 2015 Oct 14. No abstract available. PMID 26462668
- [Background] Azad MB, Sharma AK, de Souza RJ, Dolinsky VW, Becker AB, Mandhane PJ, Turvey SE, Subbarao P, Lefebvre DL, Sears MR; Canadian Healthy Infant Longitudinal Development Study Investigators. Association Between Artificially Sweetened Beverage Consumption During Pregnancy and Infant Body Mass Index. JAMA Pediatr. 2016 Jul 1;170(7):662-70. doi: 10.1001/jamapediatrics.2016.0301. PMID 27159792
- [Background] Mennella JA. Ontogeny of taste preferences: basic biology and implications for health. Am J Clin Nutr. 2014 Mar;99(3):704S-11S. doi: 10.3945/ajcn.113.067694. Epub 2014 Jan 22. PMID 24452237
- [Background] Joseph PV, Reed DR, Mennella JA. Individual Differences Among Children in Sucrose Detection Thresholds: Relationship With Age, Gender, and Bitter Taste Genotype. Nurs Res. 2016 Jan-Feb;65(1):3-12. doi: 10.1097/NNR.0000000000000138. PMID 26633761
- See also: New food labelling law in Chile — http://www.minsal.cl/reglamento-de-la-ley-de-etiquetado-de-alimentos-descarga/